CLINICAL TRIAL: NCT02118272
Title: A Multicentre, Prospective Clinical Study Evaluating the Outcomes of a New Knee System with a Physiological Rollback Mechanism
Brief Title: Clinical Study Evaluating the Outcomes of a New Knee System with a Physiological Rollback Mechanism
Acronym: K-06
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study concluded as per protocol
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-06 Physica KR
Record Dates: First submitted 2014-04-11; First posted 2014-04-21 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Primary Total Knee Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Physica KR (Other)
  Interventions: Device: Physica KR

INTERVENTIONS:
Device: Physica KR

SUMMARY:
The aim of this study is to assess the clinical, radiographic and patient-reported outcome measures (PROMs) after total knee replacement with Physica KR, define the survivorship of the implants and identify possible risk factors that may lead to failure.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females
2. Age 22-80 years
3. Any race
4. Ambulatory patients
5. Patients who have a medical condition with over 5 years of life expectancy
6. Patients requiring knee prosthesis, suitable for the use of Physica KR
7. Patients with painful primary knee osteoarthritis
8. Patients with painful secondary knee osteoarthritis
9. Patients who are suffering from inflammatory arthritis (e.g. rheumatoid arthritis)
10. Patients who have undamaged and functional collateral and posterior cruciate ligaments
11. Patients with a flexion greater than or equal to 90° on the affected side
12. Patients with a fixed flexion contracture less than 10°
13. Patients who understand the conditions of the study and are willing and able to comply with the prescribed rehabilitation and to perform all scheduled follow-up visits
14. Patients who have signed the Ethics Committee approved study-specific Informed Consent Form prior to the surgery

Exclusion Criteria:

1. Obese patients with BMI above 35 kg/m2 (severe obesity)
2. Previous partial knee replacement (unilateral, bicompartimental or patellofemoral joint replacement), patellectomy, high tibial osteotomy or femoral osteotomy in the affected knee
3. Primary Total Knee Replacement (TKR) in the affected knee
4. Varus or Valgus deformity greater than 20°
5. Patients with a fixed flexion contracture greater than 10°
6. Previous knee replacement on the contralateral side within the last year and whose outcome is achieving an KSS< 70 points
7. Patients with symptomatic OA of the hips, spine, ankles, if it can interfere with the evaluation of the target knee
8. Patients with active or any suspected infection (on the affected knee or systemic)
9. Muscular insufficiency or absence of muscoligamentous supporting structures required for adequate soft tissue balance
10. Patients with known or suspicious metal hypersensitivity
11. Recurrent medical history of severe allergic or immune-mediated reactions
12. Vascular insufficiency of lower limbs severe enough to interfere with the study evaluation
13. Current treatment or treatment within the previous 2 years before the screening visit for malignant and life-threatening non-malignant disorders
14. Any clinically significant pathology based on clinical history that the Investigator feels may affect the study evaluation
15. Any intercurrent chronic disease or condition that may interfere with the completion of the 5-year follow-up, such as liver disease, severe coronary disease, alcohol or drug abuse, disordered mental state, or other clinically significant condition
16. Patients who have significant neurological or musculoskeletal disorders or disease that may adversely affect gait and compromise functional recovery and evaluation
17. Patients who have neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device
18. Patients with systemic or metabolic disorders leading to progressive bone deterioration
19. Patients who have a medical condition with less 5 years of life expectancy
20. Previous organ transplant surgery
21. Any psychiatric illness that would prevent comprehension of the details and nature of the study
22. Participation in any experimental drug/device study within the 6 months prior to the screening visit
23. Female patients who are pregnant, nursing, or planning a pregnancy

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Knee Society Clinical Rating System (KSS) | From baseline to 5 year follow up

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | From baseline to 5 year follow-up
Oxford Knee Score (OKS) | From baseline to 5 year follow-up
Satisfaction Visual Analogue Scale (VAS) | From baseline to 5 year follow-up
Survival rate of the implant | at 3 and 5 year follow-up
Incidence of AE/SAE, ADE/SADE | From baseline to 5 year follow-up
Forgotten Joint score (FJS) | From baseline to 5 year follow-up

CONTACTS AND LOCATIONS:
Locations (3):
- Azienda Ospedaliero-universitaria Careggi, Florence, Florence, Italy
- United Kingdom (2):
  - The Royal Bournemouth Hospital, NHS Foundation Trust, Bournemouth, Dorset
  - Dorset County Hospital NHS Foundation Trust, Dorchester, Dorset

IPD SHARING:
Plan to Share IPD: No